CLINICAL TRIAL: NCT06231524
Title: Development and Validation of a AI Prognostic Model Based on DNA Ploidy, Stroma, and Nucleotyping for Synchronous Peritoneal Metastasis From Colorectal Cancer
Brief Title: Development and Validation of a PSN-AI Prediction Model
Acronym: PSN-AI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: PSN2023
Record Dates: First submitted 2024-01-04; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer; Peritoneal Metastases
Keywords: Colorectal Cancer; Synchronous peritoneal metastasis; DNA ploidy; Stroma-tumor fraction; Nucleotyping
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Primary tumor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validation cohort: A cohort of consecutive patients from the Sixth Affiliated Hospital of Sun Yat-sen University is used for model validation.
  Interventions: Other: Analyse pathologic slides

INTERVENTIONS:
Other: Analyse pathologic slides — HE-stained whole slide images were used for the validation of the PSN-AI model.

SUMMARY:
Heterogeneity concerning survival in synchronous peritoneal metastasis from patients with colorectal cancer exists, thereby further classification is urgently required. This study aimed to validate a PSN-AI model based on DNA ploidy, stroma-tumor fraction, and nucleotyping (PSN) for the prediction of survival of synchronous peritoneal metastasis from colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of synchronous peritoneal metastases of a nonappendiceal colorectal adenocarcinoma.
* Resectable disease determined by computed tomography (CT) and a peritoneal cancer index (PCI) of ≤20 at diagnostic laparoscopy or laparotomy;
* No evidence of systemic (e.g. liver, lung) colorectal metastases within three months prior to enrolment;
* Undergoing cytoreduction surgery for synchronous peritoneal metastasis from colorectal cancer.

Exclusion Criteria:

* Combined with other types of malignant tumors.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent cytoreduction surgery for synchronous peritoneal metastasis from colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At least 1-year follow up
  The time between the date of diagnosis and the date of death (due to any cause) or the date of last follow-up.

SECONDARY OUTCOMES:
Progression-free survival | At least 1-year follow up
  The time from diagnosis to the onset of disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided